CLINICAL TRIAL: NCT02562157
Title: Gastroenteric Anastomosis With Natural Orifice Translumenal Endoscopic Surgery (NOTES) Using the New Fashionned Tissue Apposing Stent Axios® for the Treatment of Antro-pyloric or Duodenal Obstructions : Prospective Evaluation of Feasibility, Efficacy and Tolerance.
Brief Title: Endoscopic Gastroenteric Anastomosis With New Tissue Apposing Stent in the Management of Antro-pyloroduodenal Obstruction : Evaluation of Feasibility, Efficacy and Tolerance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-32
Record Dates: First submitted 2015-09-17; First posted 2015-09-29 (Estimated); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Antro-pyloric and/or Duodenal Benign or Malignant Obstructions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with antro duodenal obstructions (Experimental): NOTES gastroenteric anastomosis
  Interventions: Radiation: HYALURONIQUE ACIDE

INTERVENTIONS:
Radiation: HYALURONIQUE ACIDE — Intradermal delivery of fractional CO2 laser-assisted hyaluronic acid in facial skin contouring

SUMMARY:
Achieving gastro-jejunal or duodenal anastomosis (GJA ) by exclusive endoscopically is a real goal for many years in the development and research of the transluminal endoscopic surgery (N.O.T.E.S). Endoscopic treatment, including palliative antro duodenal stenosis by metallic stent, although minimally invasive, causes problems in long-term secondary obstruction and migration. Surgical treatment of these strictures is associated with significant morbidity and mortality . The complication rate and severity of post-operative surgery after gastric bypass Roux-en-Y anastomosis or gastroduodenal fistulas remain close to 5% with a mortality of 1%. After 3 years of experimental research on porcine model, our team has developed a procedure of gastro duodenal anastomosis using transgastric endoscopic minimally invasive surgical technique (or NOTES) - LBA UMRT24 CERC laboratory , Aix-Marseille University , Faculty of Medicine North, with the aim to offer a credible alternative to conventional surgery.

Thus the investigators propose to conduct a pilot prospective intervenionnal study. The investigators hypothetized that this technique would reduce morbidity and mortality clinical but also economic consequences of surgery while making it possible to obtain excellent results permeability and long-term functionality. This method uses a new concept of tissue apposition with a fully covered metallic stent to create the anastomosis under endoscopy exclusively. Ten patients with antro duodenal obstructions requiring surgical or endoscopic bypass will be included as part of an interventional biomedical research that will be conducted in one expert center. The duration of the inclusions will be 18 months. Then, the stent will be removed three months after insertion, at the end of the healing process, and each patient will be followed for one year. The primary endpoint will be the assessment of the feasibility of the procedure for gastro duodenal anastomosis using tissue apposition stenting and NOTES in human being. The secondary endpoints will be the clinical efficacy, the long term (1 year) patency of the anastomosis, the procedure duration, adverse events, morbidity and mortality, the quality of life and the length of stay.

In case of failure of the NOTES procedure, the patient will be treated either by surgery or by conventional endoscopy according to the usual techniques without loss of chance. The risk / benefit ratio appears positive and a safety report will be issued after the first 4 inclusions. There will be no supplementary examination in patient follow-up in this study for which a CT iconography and biology are enough. The material used in the context of this work is consistent with the legislation on medical devices and has received CE Mark (tissue apposition fully covered stent Axios ®).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Benign or malignant antropyloric or duodenal obstruction leaving free the 3rd and the 4th duodenum, confirmed by CT scan or endoscopy
* Patient having been hospitalized at least once for this indication, with failure of medical treatment and/or failure or impossibility of endoscopic treatment using metallic duodenal stenting.
* Patients having under nutrition with a weight loss > 10%
* Theorical indication of surgical gastroenteric anastomosis with operating contraindication or refusal of the surgery by the patient
* Indication validated during multidisciplinary meeting
* GOOSS score = 0 or 1
* Patient having received clear and complete information and given written consent
* Patient having medical care insurrance

Exclusion Criteria:

* Contraindication to general anesthesia
* Severe hemostasis and coagulation troubles : Prothrombin level < 50% and/or platelets level < 50G/l
* History of duodenal or gastric surgery
* Pregnancy or population of vulnerable patients
* Mental deficiency
* Voluntary withdrawal of informed consent
* Discontinuation by decision of the investigator or the promotor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Feasibility of the gastroenteric anastomosis | End of procedure (up to 2 hours)
  Technical feasibility of the anstomosis endoscopically confirmed by the ability to perform the proceudre exclusively by endoscopy, and by opacification under contrast showing the patency and the absence of fistula.

SECONDARY OUTCOMES:
Clinical efficacy | 5 days to 6 months
  GOOSS score increasing by 2 points after 4 weeks of follow-up ; Weight gain > 10%
Long term patency | 15 days after stent removal, after 6 and 12 months
  Ability to pass an inflated 15mm balloon and a large channel gastroscope
Procedure duration | end of study (30 months)
Morbidity evaluation | few days, 30 days, and late adverse events
  Cotton classification
Evaluation of quality of life | until 12 months
  SF 36 Scale
Length of stay in hospitalization | end of last hospitalization (approximatively 18 months)
Procedure learning curve | end of study (30 months)
Mortality evaluation | up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Director, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France